CLINICAL TRIAL: NCT00767975
Title: Active Screening of Latent TB Infection, Treatment and Long Term Follow-up in Prison
Acronym: LTBI_prison
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Haung Li-Min, National Taiwan University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 200707047M; DOH-97-DC-1502 (Other Grant/Funding Number: Taiwan CDC)
Record Dates: First submitted 2008-01-10; First posted 2008-10-07 (Estimated); Last update posted 2010-11-29 (Estimated); Status verified 2010-11

CONDITIONS: Tuberculosis
MeSH Terms: conditions — Tuberculosis | interventions — Isoniazid; Random Allocation; Rifampin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 2 (No Intervention): For patients who diagnosed with LTBI, they choose to receive LTBI treatment depends on their willingness; if they choose not, then they are in no intervention arm.
- 1 (Experimental): Provided INH 6m or RMP 4 m; whether enter treatment arm is determined by patient's willingness
  Interventions: Drug: isoniazid , randomized, open label; Drug: rifampin, randomized, open label

INTERVENTIONS:
Drug: isoniazid , randomized, open label — isoniazid 300mg/tab 1 tab qd, 6 months (the other treatment arm is rifampin)
  Arms: 1
Drug: rifampin, randomized, open label — rifampin 300mg/capsule 2 caps qd, 4 months (the other treatment arm is isoniazid)
  Arms: 1

SUMMARY:
LTBI Treatment is effective in prison

DETAILED DESCRIPTION:
LTBI treatment will be conducted in a prison with either isoniazid or rifampin

ELIGIBILITY:
Inclusion Criteria:

* all people who is LTBI, and have ability to sign the informed concent

Exclusion Criteria:

* previously adverse effect from anti-TB medication complete treatment of TB in the pass; active TB AST, ALT > 3 times of normal limit platelet < 150 k/mm3 T-bil > 2 times of normal limit

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2384 (Actual)
Dates: Start 2008-01; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
COMPLETE RATE OF LTBI TREATMENT | 1.5 year

SECONDARY OUTCOMES:
Efficacy | 3 year

CONTACTS AND LOCATIONS:
Overall Officials: Li-Min Huang, MD, PHD, Principal Investigator — National University Hospital, Singapore
Locations (1):
- Taipei Prison, Taoyuan District, Taiwan

REFERENCES:
- [Derived] Chan PC, Yang CH, Chang LY, Wang KF, Lu BY, Lu CY, Shao PL, Hsueh PR, Fang CT, Huang LM. Latent tuberculosis infection treatment for prison inmates: a randomised controlled trial. Int J Tuberc Lung Dis. 2012 May;16(5):633-8. doi: 10.5588/ijtld.11.0504. Epub 2012 Mar 8. PMID 22410137